CLINICAL TRIAL: NCT01588067
Title: Effectiveness of Medical Therapy, Endovascular Therapy, and Surgery for Peripheral Arterial Disease.
Acronym: PAD
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CO-10-1488
Record Dates: First submitted 2012-04-04; First posted 2012-04-30 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Medical: Patients treated for PAD medically or with exercise therapy
- Endovascular: Patients with PAD treated with endovascular therapy
- Surgery: Patients with PAD treated with surgery

SUMMARY:
This study is designed to develop a clinical registry of Peripheral Arterial Disease (PAD) patients undergoing lower extremity revascularization to describe the population and assess comparative effectiveness of endovascular therapy versus surgery. In addition, this study will conduct a prospective cohort study of patients treated medically or undergoing lower extremity revascularization at the VA and Kaiser Colorado to compare changes in health status.

DETAILED DESCRIPTION:
Using electronic medical records, a registry of patients undergoing lower extremity revascularization therapy will be identified. Chart reviews with be done by an expert panel.

The prospective cohort study will ask participants to complete health status surveys before they begin therapy for PAD and again 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* presents with PAD,
* > 18 years of age,
* can complete a questionnaire, and
* has either had a change in PAD lower extremity intervention or start of a new intervention (surgical, endovascular, or medical therapy (cilostazol or exercise regimen)

Exclusion Criteria:

* dementia,
* inability to consent,
* pregnancy,
* limited life expectancy (< 6 months),
* previous endovascular or surgical revascularization within the previous 12 months,
* non English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with PAD
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Health Status at 6 months | Baseline (pre procedure), 6 months
  Health Status will be measured at baseline and six months following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Magid, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - VA Eastern Colorado Health Care System, Denver, Colorado
  - Kaiser Permanente Colorado, Denver, Colorado